CLINICAL TRIAL: NCT02350426
Title: An Adaptive Design Open Label Pilot Study in Rheumatoid Arthritis Patients to Assess Inflammation Using Molecular Imaging Techniques
Brief Title: A Study to Assess Inflammation in Rheumatoid Arthritis Using Molecular Imaging Techniques
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A decision to stop the study was made by the site and GSK project team based on pre-defined stopping criteria in the protocol
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 201659
Record Dates: First submitted 2014-12-15; First posted 2015-01-29 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — gadobutrol; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): As per randomization schedule, subjects will undergo two half body PET/CT scans (PET/CT1 and PET/CT2). During visit 1 subject will undergo PET/CT1 scan with 18F-FDG followed by PET/CT2 scan with 18F-GE-180 in visit 2. A sub-group of patients will participate in an additional dynamic PET/CT scan with 18F-GE-180 prior to their 18F-GE-180 PET/CT half body scan.
  Interventions: Other: Gadobutrol; Other: 18F-FDG; Other: 18F-GE-180
- Arm 2 (Experimental): As per randomization schedule, , subjects will undergo two half body PET/CT scans (PET/CT1 and PET/CT2). During visit 1 subject will undergo PET/CT1 scan with 18F-GE-180 followed by PET/CT2 scan with 18F-FDG in visit 2. A sub-group of patients will participate in an additional dynamic PET/CT scan with 18F-GE-180 prior to their 18F-GE-180 PET/CT half body scan.
  Interventions: Other: Gadobutrol; Other: 18F-FDG; Other: 18F-GE-180

INTERVENTIONS:
Other: Gadobutrol — Gadobutrol is a solution for intravenous (IV) injection in prefilled syringe/cartridge with a unit dose strength of 1.0 millimole (mmol)/mL solution, and will be administered at up to 0.1mmol/kg.
Other: 18F-FDG — 18F-FDG is a solution for IV injection in multidose vial, maximum 10 mL with unit dose strength of 160 megabecquerel (MBq) at maximum.
Other: 18F-GE-180 — 18F-GE-180 solution for IV injection in 10mL glass vial. Patients will receive a maximum activity of 195 MBq in a maximum volume of 10 mL (bolus) of 18F-GE-180, containing not more than 2 microgram (mcg)/mL 18F-GE-180 (20 mcg for a 10 mL dose).

SUMMARY:
This is an adaptive Positron Emission Tomography/ Computed Tomography (PET/CT) and Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI) open-label study design for the investigation of inflammation in adult rheumatoid arthritis (RA) patients, not involving therapeutic intervention. Each study participant will undergo two half body PET/CT scans from the pelvis to the bottom of the feet (including hands and wrists) with an additional bed position centred on the shoulders. One scan will be conducted with 18F-FDG and the other with 18F-GE-180. The first PET/CT scan (PET1) will be performed 4 weeks (28 +/- 2 days) after the first screening visit, whereas the second PET/CT scan (PET2) will be carried out within 2 weeks (7 +/- 7 days) after PET1. The order of PET/CT scans for each subject will be based on a computer generated randomisation schedule after the screening visit. A sub-group of study participants will be invited to undergo an additional dynamic 18F-GE-180 PET scan of a selected joint (knee or wrist) prior to their 18F-GE-180 PET/CT half body scan. The primary objective of the study is to quantify inflammation in joints of RA patients by determining 18F-FDG and 18F-GE-180 uptake using PET, and DCE-MRI parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be aged between 30 and 85 years inclusive at the time of signing the consent form.
* Stable, moderate to severe RA, based on either the 1987 American College of Rheumatology definition or the 2010 American College of Rheumatology/ European league Against Rheumatism (ACR/EULAR) classification criteria for RA (functional classes II and II).
* Disease activity score (DAS)28-erythrocyte sedimentation rate >3.2 at screening.
* Patients with at least one painful and swollen wrist or knee joint as assessed by a rheumatologist.
* Male subjects are eligible for enrolment in the study OR female subjects of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy (for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records) or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international unit per milliliter (MIU/mL) and estradiol <40 picogram/mL (pg/mL) (<147 picomole per liter [pmol/L]) is confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use two of the contraception methods listed in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method OR female subjects of child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotropin (hCG) test at screening and 4-7 days prior to dosing and agrees to use two different contraception methods listed in the protocol. Use must be established a minimum of 1 month prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception from at least one month prior to the first dose through to follow up. Contraception requirements do not apply to women with only same-sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis.
* Subjects must be capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Subjects who meet diagnostic criteria for any other rheumatic disease (e.g., lupus erythematosus).
* Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac (including ischemic heart disease), neurological, or cerebral disease, or other medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude.
* Patients not on stable medication for RA for at least 4 weeks prior to screening.
* Subjects receiving treatment with biologics will not be eligible for inclusion.
* Subjects exceeding 159 kilogram (kg) body weight.
* Subjects exceeding 195 centimeter (cm) in height.
* History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study procedures or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subjects with creatinine clearance levels <60 milliliter per minute (mL/min).
* A positive pre-study alcohol screen (alcohol breath test).
* Pregnant females as determined by positive serum HCG test at screening or prior to imaging-related procedures.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* Exposure to more than four new chemical entities within 12 months prior to the first imaging-related procedures.
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden (a significant radiation burden being defined as 10 milliSievert [mSv] in addition to natural background radiation, in the previous 3 years including the dose from this study).
* History of, or suffers from, claustrophobia or feel that they will be unable to lie still in the PET or MRI scanner for a period of 1-2 hours or fit in the PET or MRI scanner due to body size.
* Contraindication to MRI scanning (as assessed by local MRI safety questionnaire) which includes, but is not limited to, intracranial aneurysm clips or other metallic objects, history of intra-orbital metal fragments that have not been removed by a medical doctor MD), presence of a cardiac pacemaker, non-magnetic resonance (MR) compatible heart valves or other electronic device or ferromagnetic metal foreign bodies, inner ear implants or history of cancer in first degree relatives diagnosed before age of 55.
* Presence of Ala147Thr polymorphism in translocator protein (TSPO) (which confers low affinity binding of 18F-GE-180) following confirmation by genotyping assay.
* Subjects receiving treatment with Disulfiram.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-10-26 (Actual)

PRIMARY OUTCOMES:
Evaluator's assessment of image quality and potential to define abnormality | Week 8
  Half body and shoulder images from 18F-FDG and 18F-GE-180 will be visually inspected by two nuclear medicine physicians with respect to the clarity and ease of identifying abnormal high uptake in joints suspected to have inflammation. A subjective scale of abnormality will be applied to each image as follows: 3 = excellent quality; 2 = intermediate quality; 1 = poor quality but still interpretable; 0 = poor quality, not interpretable.
Standardised Uptake Value (SUV) of 18F-FDG and 18F-GE-180 | Week 8
  SUV will be derived from PET static imaging for 18F-FDG and 18F-GE-180 in selected joints. Using normalisation by weight and body surface area, SUVmax, SUVpeak and SUVmean (average of voxel values above a 75% iso-contour of SUVmax) will be calculated within the joint volume.
Tissue-to-reference Ratio (TR) of 18F-FDG and 18F-GE-180 | Week 8
  TR will be derived from PET static imaging for 18F-FDG and 18F-GE-180 in selected joints. TR will be determined using the mean image value within each joint volume, and either the blood concentration decay-corrected to the start of the PET acquisition or the mean image value within non-inflamed muscle as reference.
Total Inflammatory Volume (TIV) of 18F-FDG and 18F-GE-180 | Week 8
  TIV will be derived from PET static imaging for 18F-FDG and 18F-GE-180 in selected joints.
Exchange Rate (Ktrans) | Week 8
  Ktrans will be derived from DCE-MRI in selected joints
Interstitial Volume (Ve) | Week 8
  Ve will be derived from DCE-MRI in selected joints
Initial Rate of Enhancement (IRE) | Week 8
  IRE will be derived from DCE-MRI in selected joints
Maximal Signal Intensity Enhancement (ME) | Week 8
  ME will be derived from DCE-MRI in selected joints

SECONDARY OUTCOMES:
Visual assessment of static 18F-FDG and 18F-GE-180 images using a 4-point visual analysis scale and abnormal joint counts | Week 8
  18F-FDG and 18F-GE-180 static images will be evaluated by experienced observers with respect to the ease of identifying high uptake in joints suspected to have inflammation. Images will be assessed on the basis of a 4-point visual scale of abnormality/discernibility (0=poor quality - 4=excellent quality) and the number of abnormal joints will be counted.
PET static imaging parameters (SUV, TR and TIV) of 18F-FDG and 18F-GE-180 in selected joints | Week 8
  The correlation between PET static imaging parameters (SUV, TR and TIV) of 18F-FDG and 18F-GE-180 will be determined
18F-GE-180 radio-PK modelling indices (total distribution volume; VT) and 18F-GE-180 static imaging metrics (SUV, TR and TIV) | Week 8
  In order to verify static imaging parameters for scans, the pharmacokinetic profile of 18F-GE-180 will be determined, using dynamic PET scanning, blood sampling and HPLC analysis in a sub-cohort of RA study patients. 18F-GE-180 radio-PK parameters will be correlated with 18F-GE-180 static imaging metrics (SUV, TR and TIV)
Adverse events (AEs) and serious adverse events (SAEs) assessment | Week 8
  Number of AEs and SAEs as a measure of safety and tolerability of 18F-GE-180 and 18F-FDG

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Cambridge